CLINICAL TRIAL: NCT02095522
Title: Does COlchicine Improve EnDothElial Function in Non ST Elevation Myocardial Infarction Patients?: A Prospective Randomized, Double-blind Placebo Controlled Study
Brief Title: COlchicine Improve EnDothElial Function in Non ST Elevation Myocardial Infarction Patients
Acronym: CODEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators did not find suiable patients
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, michal roll, Tel-Aviv Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-13-YA-0636-CTIL
Record Dates: First submitted 2014-03-06; First posted 2014-03-24 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: NSTEMI
Keywords: colchicine NSTEMI endothelial function inflammation
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine 1mg per day for one month
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo 1mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 1mg per day for one month
  Arms: Colchicine
Drug: Placebo — Placebo
  Other Names: Placebo tablet 1mg per day for a month
  Arms: Placebo

SUMMARY:
Colchicine has antiinflammatory properties. It has been shown to be effective in improving outcome in stable coronary disease. The exact mechanism is unclear. Study objective: to assess the effect of colchicine on endothelial function using the EndoPAT™ in NSTEMI Patients.

Study Hypothesis: There will be a significant difference on the RH-PAT levels of the patients who were in treated with colchicine versus the placebo group Study design and patient Selection One hundred and forty patients with the diagnosis of Non ST Elevation Myocardial Infarction will be enrolled to a prospective randomized double-blind placebo controlled study in Tel Aviv Medical Center, Tel Aviv, Israel. Patients will be recruited during their hospitalization before cardiac catheterization. All patients will sign an informed consent.

Primary outcome will be the improvement in endothelial function between baseline and after 1 month in both groups

DETAILED DESCRIPTION:
Study design and patient Selection One hundred and forty patients with the diagnosis of Non ST Elevation Myocardial Infarction (NSTEMI) will be enrolled to a prospective randomized double-blind placebo controlled study in Tel Aviv Medical Center, Tel Aviv, Israel. Patients will be recruited during their hospitalization before cardiac catheterization. All patients will sign an inform consent. Study will be published on NIH clinicaltrials.com database.

Inclusion and exclusion criteria are presented in Table 1 Table 1: Patient Selection Inclusion criteria

1. NSTEMI Diagnosis 2. Patients above the age of 18 3. Informed consent Exclusion criteria

1. Hemodynamic instability
2. Pregnant women
3. Peripheral vascular disease with feeble or absent peripheral pulses
4. Restlessness and/or chaotic breathing
5. Renal dialysis
6. Severe aortic valve insufficiency/Stenosis
7. Severe mitral valve insufficiency
8. Congenital cardiac malformations (structural heart diseases)
9. Known extra-cardiac shunts
10. Major surgery within 30 days
11. Any medical condition that would impair participation (e.g. progressive neurological disorders, mental illness)
12. Known intolerance to colchicine
13. Ejection fraction less than 35% or past admission for CHF exacerbation in the last 30 days.
14. Inflammatory diseases
15. Current treatment with steroids, NSAID, chemotherapy or biologic medications

Pre Study exam

After enrollment, patients will undergo the following baseline procedure:

1. Physical examination and medical interview
2. Endothelial function using the EndoPat® before planned cardiac catheterization
3. Blood tests- see below for description

Blood sampling An 18-gauge cannula will be placed in an antecubital vein for blood sampling. Blood sample analyses will be performed using reagents, calibrators and control materials from Bayer Diagnostics (Berkshire, England) on the ADVIA 1650. A 40 ml blood sample will be obtained as described below. Blood tests timing is detailed at the end in the flow chart.

Each Patient will provide 40ml of blood for the following blood tests

1. Full chemistry including: lipid levels, thyroid function, liver enzymes function, Troponin, CPK, HbA1c, uric acid, and glucose levels.
2. Blood count
3. Inflammatory biomarker (hs-CRP, fibrinogen, IL-6, IL-1B, IL-18, MMP, Lp-PLA2, procalcitonin, IL-10, IL-35, TNFa, AchE, , PAI-1, MPO, cholinergic status. etc.)
4. Endothelial function markers: Endothelin-1, I-CAM, V-CAM, superoxide dismutase ADMA, and oxidized LDL
5. Serum Samples will be stored for future testing.

PAT score:

Peripheral arterial tonometry signals will be obtained using the EndoPAT 2000 device (Itamar Medical Inc., Caesarea, Israel), which has been validated and used previously to assess peripheral arterial tone in other populations. 14-17 Briefly, EndoPAT bio-sensors are placed on the index fingers of both arms. EndoPAT quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard blood pressure cuff). When the cuff is released, the surge of blood flow causes an endothelium-dependent Flow Mediated Dilatation (FMD). The dilatation, manifested as reactive hyperemia, is captured by EndoPAT as an increase in the PAT Signal amplitude. A post-occlusion to pre-occlusion ratio is calculated by the EndoPAT software, providing the EndoPAT index. In addition, the EndoPAT system will measure heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

1. NSTEMI Diagnosis
2. Patients above the age of 18
3. Informed consent

Exclusion Criteria:

1. Hemodynamic instability
2. Pregnant women
3. Peripheral vascular disease with feeble or absent peripheral pulses
4. Restlessness and/or chaotic breathing
5. Renal dialysis
6. Severe aortic valve insufficiency/Stenosis
7. Severe mitral valve insufficiency
8. Congenital cardiac malformations (structural heart diseases)
9. Known extra-cardiac shunts
10. Major surgery within 30 days
11. Any medical condition that would impair participation (e.g. progressive neurological disorders, mental illness)
12. Known intolerance to colchicine
13. Ejection fraction less than 35% or past admission for CHF exacerbation in the last 30 days.
14. Inflammatory diseases
15. Current treatment with steroids, NSAID, chemotherapy or biologic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Improvement of RH-PAT at 1 month (a marker of endothelial function) | 1 month
  RH-PAT will be measured before the angiography and after one month.

SECONDARY OUTCOMES:
Improvement in inflammatory biomarkers (before cardiac catheterization, after cardiac catheterization and at 1 month time follow-up) | 1 month
  biomarkers will be assessed before and after the angiography. Comparison of the biomarker levels will be assessed between the two treatment groups
Improvement in endothelial function markers. | 1 month
  serum ICAM VACAM and endothelin will be measured
inflammatory biomarkers Improvement of heart rate variability (HRV) | 1 month
Changes in cholinergic status | 1 month
  serum ACHE will be measured at randomization and after one month
Reduction of Acute Kidney Injury post PCI | 1 month
  AKI will be defined per AKIN as an increase of 0.3mg/dl. The two treatment groups will be compared
Reduction in radial artery occlusion | acute
Reduction of peri-procedural myocardial infarction | 1 month
Major adverse clinical events (MACE) defined as a composite of all-cause mortality, myocardial infarction, repeat revascularization, and 30 day readmission rate | 1 month
quality of life under colchicine treatment | 1 month
  The investigators will assess this outcome using a standard quality of life questionnaire (EQ5).
Safety | up to 1 year
  Safety will be assessed by comparing adverse events between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Arbel, MD, Principal Investigator — Tel Aviv Medical Center
Locations (2):
- Israel (2):
  - Tel Aviv Medical Center, Tel Aviv, Israel
  - Sourasky medical center (Ichilov), Tel Aviv

IPD SHARING:
Plan to Share IPD: No